CLINICAL TRIAL: NCT04226131
Title: MusculRA: The Effects of Rheumatoid Arthritis on Skeletal Muscle Biomechanics
Acronym: MusculRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00103552
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Rheumatoid Arthritis; Healthy Controls
Keywords: Skeletal Muscle
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection; Restraint, Physical; Spectroscopy, Near-Infrared; Body Composition; Exercise Test; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: 15 participants with early RA defined as duration of disease/symptoms of less than 6 months (where "duration" denotes the length of time the patient has had symptoms/disease, not the length of time since RA diagnosis) AND prior to starting biologic DMARD therapy and 15 age-, sex-, and BMI-matched controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Rheumatoid Arthritis (RA) (Other): Early RA defined as duration of disease/symptoms of less than 6 months (where "duration" denotes the length of time the patient has had symptoms/disease, not the length of time since RA diagnosis) AND prior to starting biologic Disease-modifying anti-rheumatic drugs (bDMARD) therapy
  Interventions: Other: Blood Draw; Other: Disease Activity (DAS-28) Assessment; Other: Skeletal Muscle Mitochondrial Respiratory Capacity; Other: Muscle Biopsy; Other: Body Composition; Other: Cardiopulmonary Exercise Test (CPET); Other: Strength Testing; Other: Questionnaires; Other: Skeletal Muscle Biomechanical Property Assessment
- Age-, Sex-, BMI-matched Healthy Controls (Other): Healthy Controls.
  Interventions: Other: Blood Draw; Other: Skeletal Muscle Mitochondrial Respiratory Capacity; Other: Muscle Biopsy; Other: Body Composition; Other: Cardiopulmonary Exercise Test (CPET); Other: Strength Testing; Other: Questionnaires; Other: Skeletal Muscle Biomechanical Property Assessment

INTERVENTIONS:
Other: Blood Draw — A study nurse will draw up to 150 mL of blood to measure erythrocyte sedimentation rate (ESR) and measures of immune cell function. ESR is a common hematology test that is a measure of inflammation.
Other: Disease Activity (DAS-28) Assessment — Participants in the RA cohort will receive a 28-joint examination by the study physician to assess RA disease activity and report their overall health assessment.
  Arms: Early Rheumatoid Arthritis (RA)
Other: Skeletal Muscle Mitochondrial Respiratory Capacity — Near-Infrared Spectroscopy (NIRS) will be used to measure oxidative capacity of forearm flexor digitorum profundus and medial gastrocnemius muscles using the PortaMon device (Artinis Medical Systems, The Netherlands). NIRS is a low-cost, non-invasive method that estimates muscle oxidative capacity by measuring oxygen consumption (mVO2) recovery kinetics via assessment of intramuscular oxy- and deoxy-hemoglobin concentration following a sequence of brief, rapid arterial cuff occlusions. NIRS measures mitochondrial oxidative function as the mVO2 recovery rate constant k. In the absence of blood flow, changes in muscle oxygenation occur via oxygen consumption alone. In persons without RA, this non-invasive approach is highly correlated with muscle respiratory capacity assessed via muscle biopsies using in situ permiabilized fiber bundles and the Oroboros O2k system.
  Other Names: Near-Infrared Spectroscopy (NIRS)
Other: Muscle Biopsy — After local anesthesia (xylocaine, 2%) is injected, a small incision will be made in the thigh. Four to six small pieces of muscle about the size of a pea will be surgically removed. The incision site will be closed using steri-strips and/or derma-bond, and a light dressing applied.
Other: Body Composition — Body composition assessments include circumference measurements and the BOD POD®. Minimal waist circumference measurements will be taken using a tape measure.
Other: Cardiopulmonary Exercise Test (CPET) — Cardiorespiratory aerobic capacity (VO2 peak), will be assessed using a maximal treadmill test protocol with cardiopulmonary gas exchange. Subjects will be asked to exercise on a treadmill to their perceived maximum ability and effort during which time they will have a mouthpiece in their mouth to determine maximal oxygen use/consumption through breathing. For safety purposes the subject will be monitored by electrocardiogram (ECG) and their blood pressure will be measured at rest and throughout the exercise phase of this test.
Other: Strength Testing — Strength assessments will include dynamometry-assessed grip and quadriceps strength (Cybex HUMAC NORM, Comp Sports Med, Inc., Stoughton, MA) tests
Other: Questionnaires — Measures include global health, pain, fatigue, physical function, self-efficacy for disease management and sleep.
Other: Skeletal Muscle Biomechanical Property Assessment — Passive skeletal muscle stiffness and elasticity measurements of bilateral biceps brachii, flexor carpi radialis, vastus lateralis, and tibialis anterior using mechanical deformation with myotonometry using the MyotonPro device.
  Other Names: Myotonometry

SUMMARY:
Persons with rheumatoid arthritis (RA) suffer from increased disability and mortality, in part resulting from skeletal muscle impairments. In this study, our objective is to determine if skeletal muscle biomechanical properties are altered in RA. Up to 15 participants with early RA defined as duration of disease/symptoms of less than 6 months (where "duration" denotes the length of time the patient has had symptoms/disease, not the length of time since RA diagnosis) AND prior to starting biologic Disease-modifying anti-rheumatic drugs (bDMARD) therapy and 15 age-, sex-, and BMI-matched controls will undergo clinical assessments of skeletal muscle stiffness and elasticity as measured by the hand-held MyotonPro device. Additional study participant assessments include cardiopulmonary exercise testing, muscle strength testing, body composition measurement using BodPod, muscle oxidative capacity testing using near-infrared spectroscopy, and thigh muscle needle biopsies to compare clinical findings to an ex vivo cultured myobundle system. Primary statistical analyses will be comparisons of skeletal muscle parameters in RA compared to controls and correlations to determine relationships between variables. Thigh muscle biopsies are a low-risk procedure that may cause minor local soreness and bleeding; all other clinical assessments are non-invasive and will induce minimal discomfort to participants.

DETAILED DESCRIPTION:
Study design: Up to 30 adults, 25-75 yrs. of age may be recruited and enrolled to participate in a cross-sectional study. Subjects will be divided between two cohorts: 1) persons with early RA (n=15) and 2) age-, sex-, Body Mass Index (BMI)-matched healthy controls (n=15). The goal is to have equal numbers between groups complete the study. Early RA defined as duration of disease/symptoms of less than 6 months (where "duration" denotes the length of time the patient has had symptoms/disease, not the length of time since RA diagnosis) AND prior to starting biologic DMARD therapy were chosen to minimize the effect of medications on skeletal muscle.

Demographics and comorbidities will be assessed via self-report during an initial phone screening interview, with confirmation from the computerized medical record. Once it has been determined that the subject meets pre-screening criteria, they will be scheduled for Visit-1.

Phone Pre-Screening: Demographics and comorbidities will be assessed via self-report during an initial phone screening interview, with confirmation from the electronic medical record. Once it has been determined that the subject meets pre-screening criteria, they will be scheduled for a virtual study information/consent session.

Online surveys: After completion of the e-consent process, participants will be provided a REDCap survey link via email to complete some online questionnaires about their overall health, pain, fatigue, physical function, sleep and ability to manage their disease.

The study involves two on-site study visits at the Duke Center for Living; each visit lasts approximately 2.5 hours.

Study participants will undergo the following at Visit 1:

* Brief medical history including list of medications
* PROMIS Measures (If unable to complete online prior to Visit-1)
* Anthropometric Measurements: Height/Weight/Body Mass Index
* Vitals: Resting Blood Pressure and Heart Rate
* Fasting Blood Draw
* Physician RA Joint Assessment: Disease Activity (DAS-28) Assessment
* MyotonPro Skeletal Muscle Biomechanical Assessments
* NIRS Muscle Oxidative Capacity Test
* Muscle Biopsy

Brief Medical History and Medication Review: A brief medical history including list of medications will be performed by study staff.

Questionnaires: Using Duke's REDCap (Research Electronic Data Capture) interface, a battery of Patient-Reported Outcomes Measurement Information System (PROMIS) self-reported health outcome measures has been added to a computerized interface and will be associated with this investigation. Measures include global health, pain, fatigue, physical function, self-efficacy for disease management and sleep. Of note, staff testing of this battery indicated this could be completed between 10 and 12 minutes; the investigators project participants may take longer, expecting approximately 30 minutes. Except for global health, scoring is performed by the computerized REDCap interface. Specific measure names and versions as listed in REDCap are listed below:

* PROMIS SF v1.1 Global Health
* PROMIS SF v2.0 Physical Function 20a
* PROMIS Scale v1.0 Pain Intensity 3a
* PROMIS SF v1.0 General Life Satisfaction 5a
* PROMIS Bank v1.0 Short Form Fatigue 8a
* Stanford Brief Activity Survey

Study participants will undergo the following at Visit 2:

* BodPod and Minimal Waist Circumference
* Strength Tests

  * Isometric Leg Extension Machine - Quadriceps / Hamstrings Strength
  * Hand Dynamometer - Grip Strength
* Cardiopulmonary Exercise Test

ELIGIBILITY:
Inclusion Criteria: Study participants will include 25-75 year-old adults with early rheumatoid arthritis and healthy age-, gender-, and BMI-matched controls.

* Rheumatoid arthritis participants will all be seropositive (positive rheumatoid factor or anti-citrullinated protein antibody) or with erosions typical of RA on radiographs.
* Meet 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Classification Criteria for RA.
* Early RA defined as duration of disease/symptoms of less than 6 months (where "duration" denotes the length of time the patient has had symptoms/disease, not the length of time since RA diagnosis) AND prior to starting biologic DMARD therapy.
* Participants will not be engaging in regular exercise (According to 2018 US guidelines): not more than 150 minutes per week of moderate intensity exercise or 75 minutes per week of vigorous intensity exercise) for at least three months prior to consent.

Exclusion Criteria:

* Early RA participants will be excluded if they have already started bDMARD therapy.
* The investigators will exclude persons using non-aspirin anticoagulants that would complicate the biopsy. There will be a wash-out period of seven days for anti-platelet agents, and three days for NSAIDs prior to biopsies.
* Uncontrolled thyroid diseases
* Chronic obstructive lung disease
* Parkinson's disease
* Ankylosing spondylitis
* Congestive Heart Failure Class III and above will be excluded based on recognized effects on skeletal muscle.
* Patients with absolute or relative contraindications to exercise will be excluded: recent (<6 months) acute cardiac event, unstable angina, uncontrolled dysrhythmias causing symptoms or hemodynamic compromise, symptomatic aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus, acute myocarditis or pericarditis, suspected or known dissecting aneurism or acute systemic infection, left main coronary stenosis, moderate stenotic valvular heart disease, outflow tract obstruction, high degree atrioventricular (AV) block, ventricular aneurysm.
* Uncontrolled metabolic disease (e.g. diabetes, thyrotoxicosis, myxoedema)
* Uncontrolled pulmonary disease (e.g. severe COPD or pulmonary fibrosis)
* Mental or physical impairment leading to inability to exercise adequately
* Pregnant women will be excluded as determined via menstrual history/self-reporting.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Muscle stiffness and elasticity | Baseline
  Determine whether passive skeletal muscle stiffness (Newtons/meters) and elasticity (logarithmic decrement) are different in RA compared to matched healthy controls.

SECONDARY OUTCOMES:
Myobundle function | Baseline
  Determine whether myobundle function, including force production and tissue stiffness (kPa), in RA differs compared to controls.
Janus kinase/signal transducers and activators of transcription 3 pathway (JAK/STAT3) signaling in skeletal muscle | Baseline
  Determine whether JAK/STAT3 signaling is upregulated in RA skeletal muscle compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Kim M Huffman, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No